CLINICAL TRIAL: NCT03086798
Title: Comparison Techniques of Magill Forceps and Cuff Inflation to Facilitate Nasotracheal Tube Placement Under Video-laryngoscope Use
Brief Title: Comparison of Different Tools to Facilitate Nasotracheal Tube Placement Under Video-laryngoscope Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KMUHIRB-F(II)-20150058
Record Dates: First submitted 2017-02-01; First posted 2017-03-22 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2018-03

CONDITIONS: Nasotracheal Intubation
Keywords: Magill forceps; cuff inflation; Nasotracheal Intubation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magill forceps (Experimental): experimental Magill forceps group: Magill forceps technique to facilitate nasotracheal tube advancement into trachea
  Interventions: Procedure: Magill forceps
- cuff inflation (Experimental): experimental cuff inflation group: cuff inflation technique to facilitate nasotracheal tube advancement into trachea
  Interventions: Procedure: cuff inflation

INTERVENTIONS:
Procedure: Magill forceps — Magill forceps techniques to facilitate nasotracheal tube advancement into trachea
  Arms: Magill forceps
Procedure: cuff inflation — cuff inflation techniques to facilitate nasotracheal tube advancement into trachea
  Arms: cuff inflation

SUMMARY:
to investigate the effectiveness of techniques of either using Magill forceps or cuff inflation in facilitation of nasotracheal tube advancement into trachea

DETAILED DESCRIPTION:
Patients who undergo oxo-maxillofacial surgery need naso-tracheal intubation to present good surgical view-field. but, sometimes, the naso-tracheal tube is unable to advance from nasopharynx, oropharynx, into trachea without assistance. Using techniques of either Magill forceps or cuff inflation is advantageous is not determined.

ELIGIBILITY:
Inclusion Criteria:

1. patients with American Society of Anesthesiologists physical status I-III
2. aged 20-65 years
3. Requiring Nasotracheal Intubation under general anesthesia
4. unlimited mouth open
5. unlimited neck motion

Exclusion Criteria:

1. mouth open < 3 cm
2. Ankylosing arthritis patients.
3. BMI≧35 kg/m2

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
the technique spending time in this time interval and first attempt successful rate | 10 minutes
  to measure the time taken of either using Magill forceps or with cuff inflation techniques in successfully intubated patients

SECONDARY OUTCOMES:
total intubation time taken | half an hour
  measure the whole intubation time taken from tube tip into selected nostril, to nasopharynx, to oropharynx, into trachea, till capnography showing of 3 consecutive CO2 waveforms
glottic injury and cuff damages during tube advanced | half an hour
  to assess the bleeding point of glottic area and the cuff injury of endotracheal tube
postoperative nasal bleeding, sore throat and hoarseness | 2 days
  Events of intubating related nasal bleeding were measured on selected nostril and oral cavity at 3 minutes post-intubation. Incidences of sore throat and hoarseness are evaluated before patients out of recovery room and the coming morning

CONTACTS AND LOCATIONS:
Overall Officials: Kuang I Cheng, MD, PhD, Study Director — Department of anesthesiology, Kaohsiung Medical University, Taiwan
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided